CLINICAL TRIAL: NCT05488093
Title: Evaluation of Movement and Muscular Alterations in Subjects With Severe Knee Osteoarthritis Who Are to Receive a Total Knee Replacement
Brief Title: Evaluation of Mobility in Subjects With Severe Knee Osteoarthritis Who Are to Undergo Total Knee Replacement
Acronym: MOUV-GOPRO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RECHMPL22_0051
Record Dates: First submitted 2022-08-02; First posted 2022-08-04 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis; mobility; inertial sensors; sarcopenia
MeSH Terms: conditions — Osteoarthritis, Knee; Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- total knee replacement surgery group (Experimental): The study will be conducted in 4 visits:
  * a pre-inclusion visit during a routine care consultation where the patient will be informed about the study
  * a V1 inclusion visit (pre-surgery of the knee) during which informed consent, clinical examination, VAS, self-questionnaires, DXA, X-SENS sensor, MRI, isokinetism will be collected
  * a V2 visit during the operation, during which biological samples will be taken (muscle biopsy, collection of osteoarticular parts, and serum collection)
  * a V3 visit at 12 months with a clinical examination, EVA, self-questionnaires, DXA, isokinetics, X-SENS sensor, serum collection, and collection of adverse events.
  Interventions: Device: X-sens sensor

INTERVENTIONS:
Device: X-sens sensor — the procedure will include:
  * 7 to 8 sensors (Foot, leg, thigh, pelvis and chest possibly).
  * 5 movements/exercises for the patients, each exercise performed 3 times except walking
  * Analysis of 20m walking cycle (normal speed, most natural arm movement, 4 return trips of 20m):
  * Climbing up and down stairs (using the public stairs of the rheumatology access department, 6 steps of 20 cm height, at normal speed, without using the handrail)
  * Getting up from a chair without the help of hands (start standing, then the patient sits, leans and stands up, feet together, without taking the feet off the floor, using one and the same chair for each patient with a height of 50 cm)

SUMMARY:
Osteoarthritis (OA) is the most common joint disease. It is characterized by a progressive destruction of all the components of the joint, especially the cartilage. This leads to pain, loss of mobility and can be a major handicap for some patients.

Gonarthrosis, or osteoarthritis of the knee, affects 30% of people between the ages of 65 and 75 and is one of the most disabling conditions. In the final stage, the only therapeutic option to relieve patients is to replace the joint with a total knee prosthesis.

Thanks to the contribution of an evaluation technique based on inertial sensors (X-SENS device), our objective is to better evaluate and understand the movement deficit in knee OA subjects.

The hypothesis is that, thanks to the contribution of a technique based on inertial sensors (X-SENS), the investigators can better evaluate the movement deficit of knee OA subjects. The goal is to propose specific, rapid telekinetic biomarkers, allowing a better evaluation of functional improvements following therapeutic interventions, such as a total knee replacement.

DETAILED DESCRIPTION:
Osteoarthritis is the most common joint disease. It is characterized by a progressive destruction of all the components of the joint, especially the cartilage. This leads to pain, loss of mobility and can be a major disability for some patients.

Knee osteoarthritis affects 30% of people between the ages of 65 and 75 and is one of the most disabling conditions. In the final stage, the only therapeutic option to relieve patients is to replace the joint with a total knee prosthesis.

Previous research has shown that self-administered questionnaires to assess the benefits of management in knee osteoarthritis were limited and didn't accurately describe recovery from total knee replacement.

Functional performance tests can objectively capture a patient's mobility, but each test only approaches a small number of parameters involved in movement, which is not representative of the subject's experiences in daily life (walking, going up/down stairs, getting up from a chair).

In knee OA the assessment of pain and function is often based on validated parameters (visual analog scales and/or self-questionnaires) but variable over time (during the day, depending on physical activity or between 2 medical visits).

Given these challenges, there is great interest in using low-cost wearable sensors to develop mobile tools to obtain functional data on patients.

Thanks to the contribution of an evaluation technique based on inertial sensors (X-SENS device), the objective is to better evaluate and understand the movement deficit of of knee OA subjects.

The investigators believe that the combination of clinical, biological, imaging and mobility parameters will allow us to identify prognostic factors for OA.

The hypothesis is that, thanks to the contribution of a technique based on inertial sensors (X-SENS), the investigators can better evaluate the movement deficit of knee OA subjects. The goal is to propose specific, rapid telekinetic biomarkers, allowing a better evaluation of functional improvements following therapeutic interventions, such as a total knee replacement.

Another hypothesis is to better understand the alterations in mobility of the knee OA subject by studying several parameters: contractile function of the quadriceps; changes in body composition and muscle volume; and biological functions of muscle fibers and joint tissue.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 60 years old
* Presence of unilateral knee osteoarthritis (Kellgren and Lawrence radiographic stage ≥ 3) in the femorotibial compartment and/or Iwano stage ≥2 in the femoropatellar compartment);
* Average VAS (Visual Analogic Scale) pain on a reference joint (knee) > 40/100 during the past month.
* Indication for prosthetic knee surgery (total knee replacement)
* Failure of a well-conducted medical treatment (at least one prior infiltration with corticoids or hyaluronic acid or PRP (Platelet-rich plasma))

Exclusion Criteria:

* Presence of an inflammatory joint disease (rheumatoid arthritis, spondyloarthritis, microcrystalline pathology)
* Presence of a post-traumatic gonarthrosis
* Frontal deformity of the lower limb > 15
* Preoperative flessum > 15° or preoperative knee mobility < 90°
* Neurological pathology
* Spinal pathology that is painful or causes deformity (severe Cobb scoliosis > 20°)
* History of trauma or surgery of the lower limbs in the last two years,
* Presence of at least one lower limb prosthesis (total hip or ankle prosthesis)
* Subject with a contraindication to MRI examination (pacemaker, neurosensory stimulators, cardiac defibrillator, cochlear implants, ferromagnetic ocular or cerebral foreign bodies...)
* Subjects with a contraindication to DXA examination (coronary stent or metallic cardiac sutures, pacemaker or automatic defibrillator, obesity with a BMI > 35kg/m2, insulin pump, weight over 200kgs)
* Subject with a legal protection measure (guardianship, curatorship)
* Subject under legal protection
* Subject not affiliated to a social security system or not benefiting from such a system
* Absence of informed written consent

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-03-30 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Changes in inertial parameters before and after total knee replacement (TKR) | between baseline and 12 months
  Angular measurements in the sagittal plane during flexion and extension of the knee at 2 different times (before/after TKR) during functional movements by specifying the flexion angle at foot contact, the peak flexion angle at the beginning of the swing phase, the peak extension angle during the swing phase.
  Measurements will be taken with Xsens sensors

SECONDARY OUTCOMES:
percentage association of knee kinematics parameters with the pain VAS score at baseline | at baseline
  evaluate the percentage of association between kinematic parameters and the pain VAS score.
  the kinematic parameters of the knee are measured via the Xsens sensors
  The VAS is patient self-assessment pain scale. A high score indicates severe pain (0 = absence of pain, 100 = severe pain)
percentage association of knee kinematics parameters with the pain VAS score at 12 months | at 12 months
  evaluate the percentage of association between kinematic parameters and the VAS score.
  the kinematic parameters of the knee are measured via the Xsens sensors
  The VAS is patient self-assessment pain scale. A high score indicates severe pain (0 = absence of pain, 100 = severe pain)
percentage association of knee kinematics parameters with IPAQ score at baseline | at baseline
  evaluate the percentage of association between kinematic parameters and the IPAQ (International Physical Activity Questionnaire) score
  the kinematic parameters of the knee are measured via the Xsens sensors
  IPAQ test allows us to estimate over the last 7 days the time spent doing physical activities (intense and moderate), the time spent walking and the time spent sitting.
  By multiplying the minutes of daily activity by an activity coefficient (3.3 for walking, 4 for intense physical activity and 8 for moderate), we have a score in MET/min/week.
percentage association of knee kinematics parameters with IPAQ score at 12 months | at 12 months
  evaluate the percentage of association between kinematic parameters and the IPAQ (International Physical Activity Questionnaire) score
  the kinematic parameters of the knee are measured via the Xsens sensors
  IPAQ test allows us to estimate over the last 7 days the time spent doing physical activities (intense and moderate), the time spent walking and the time spent sitting.
  By multiplying the minutes of daily activity by an activity coefficient (3.3 for walking, 4 for intense physical activity and 8 for moderate), we have a score in MET/min/week.
percentage association of knee kinematics parameters with clinical parameters at baseline | at baseline
  evaluate the percentage of association between kinematic parameters and the actimeter
  the kinematic parameters of the knee are measured via the Xsens sensors
percentage association of knee kinematics with clinical parameters at 12 months | at 12 months
  evaluate the percentage of association between kinematic parameters and the actimeter
  the kinematic parameters of the knee are measured via the Xsens sensors
percentage association of knee kinematics parameters with KOOS score at baseline | at baseline
  evaluate the percentage of association between kinematic parameters and the KOOS (Knee Injury and Osteoarthritis Outcome Score) score
  KOOS test is a self-administered questionnaire that measures the patient's opinion of their knee health, symptoms and functionality. It contains 42 items divided into the categories of symptoms, pain, activities of daily living, sports and quality of life. The patient has 5 response modalities ranging from "not at all" to "a lot" and gives a score out of 100.
  the kinematic parameters of the knee are measured via the Xsens sensors
percentage association of knee kinematics parameters with KOOS score at 12 months | at 12 months
  evaluate the percentage of association between kinematic parameters and the KOOS (Knee Injury and Osteoarthritis Outcome Score) score
  KOOS test is a self-administered questionnaire that measures the patient's opinion of their knee health, symptoms and functionality. It contains 42 items divided into the categories of symptoms, pain, activities of daily living, sports and quality of life. The patient has 5 response modalities ranging from "not at all" to "a lot" and gives a score out of 100.
  the kinematic parameters of the knee are measured via the Xsens sensors
percentage association of knee kinematics parameters with pain detect score at baseline | at baseline
  evaluate the percentage of association between kinematic parameters and the pain detect score
  pain DETECT is used to discriminate between neuropathic and nociceptive pain. It contains 9 questions: the first 7 deal with the assessment of pain from 0 (absent) to 5 (strongly noticed), question 8 deals with the evolution of pain (from -1 to 2), and the last one deals with the presence of radiating pain (2 points if yes, 0 if no).
  A score ≤ 12 indicates that the pain is unlikely to have a neuropathic component, whereas a score ≥ 19 suggests that the pain is likely to have a neuropathic component.
  the kinematic parameters of the knee are measured via the Xsens sensors
percentage association of knee kinematics parameters with pain detect score at 12 months | at 12 months
  evaluate the percentage of association between kinematic parameters and the pain detect score
  pain DETECT is used to discriminate between neuropathic and nociceptive pain. It contains 9 questions: the first 7 deal with the assessment of pain from 0 (absent) to 5 (strongly noticed), question 8 deals with the evolution of pain (from -1 to 2), and the last one deals with the presence of radiating pain (2 points if yes, 0 if no).
  A score ≤ 12 indicates that the pain is unlikely to have a neuropathic component, whereas a score ≥ 19 suggests that the pain is likely to have a neuropathic component.
  the kinematic parameters of the knee are measured via the Xsens sensors
percentage association of knee kinematics parameters with OASIS score at baseline | at baseline
  evaluate the percentage of association between kinematic parameters and the OASIS (Overall Anxiety Severity and Impairment Scale) score
  OASIS assesses the patient's experience along 8 dimensions: sensory description, symptoms associated with arthrosis, pain rhythm, triggers, physical activity, mood, self-representation and finally general symptoms.
  the kinematic parameters of the knee are measured via the Xsens sensors
percentage association of knee kinematics parameters with OASIS score at 12months | at 12 months
  evaluate the percentage of association between kinematic parameters and the OASIS (Overall Anxiety Severity and Impairment Scale) score
  OASIS assesses the patient's experience along 8 dimensions: sensory description, symptoms associated with arthrosis, pain rhythm, triggers, physical activity, mood, self-representation and finally general symptoms.
  the kinematic parameters of the knee are measured via the Xsens sensors
percentage association of knee kinematics parameters with FJS-12 score at baseline | at baseline
  evaluate the percentage of association between kinematic parameters and the FJS-12 (Forgotten Joint Score-12) score
  FJS-12 assesses the ability of patients to forget their TKP in activities of daily living. It contains 12 items, rated from 0 (no awareness of the knee) to 4 (permanently). The score varies from 0 (extremely annoying prosthesis) to 100 (low awareness of the joint/prosthesis). This score is very relevant since it allows the practitioner to evaluate the patient's feelings about the success of the operation.
  the kinematic parameters of the knee are measured via the Xsens sensors
percentage association of knee kinematics parameters with FJS-12 score at 12 months | at months
  evaluate the percentage of association between kinematic parameters and the FJS-12 (Forgotten Joint Score-12) score
  FJS-12 assesses the ability of patients to forget their TKP in activities of daily living. It contains 12 items, rated from 0 (no awareness of the knee) to 4 (permanently). The score varies from 0 (extremely annoying prosthesis) to 100 (low awareness of the joint/prosthesis). This score is very relevant since it allows the practitioner to evaluate the patient's feelings about the success of the operation.
  the kinematic parameters of the knee are measured via the Xsens sensors
percentage association of knee kinematics parameters with MNA score at baseline | at baseline
  evaluate the percentage of association between kinematic parameters and the MNA (Mini Nutritional Assessment) score
  MNA is a 2-part questionnaire that aims to identify elderly people who are malnourished or at risk of malnutrition (from age 65).
  The first part is a 14-point screening score that assesses the patient's motor skills, weight loss, BMI and physical condition. If the patient has less than 11 points, he/she is invited to continue with the rest of the questionnaire, which looks at his/her eating habits, hydration, arm circumference, etc.
  Nutritional status is considered poor if the score is < 17/30 and "at risk of malnutrition" if the score is between 17 and 23.5.
  the kinematic parameters of the knee are measured via the Xsens sensors
percentage association of knee kinematics parameters with MNA score at 12 months | at 12 months
  evaluate the percentage of association between kinematic parameters and the MNA (Mini Nutritional Assessment) score
  MNA is a 2-part questionnaire that aims to identify elderly people who are malnourished or at risk of malnutrition (from age 65).
  The first part is a 14-point screening score that assesses the patient's motor skills, weight loss, BMI and physical condition. If the patient has less than 11 points, he/she is invited to continue with the rest of the questionnaire, which looks at his/her eating habits, hydration, arm circumference, etc.
  Nutritional status is considered poor if the score is < 17/30 and "at risk of malnutrition" if the score is between 17 and 23.5.
  the kinematic parameters of the knee are measured via the Xsens sensors
percentage association of knee kinematics parameters with SARC-F score at baseline | at baseline
  evaluate the percentage of association between kinematic parameters and the SARC-F (Strength, assistance with walking, rising from a chair, climbing stairs, and falls) score
  SARC-F is for the early detection of sarcopenia. It contains 5 questions with 3 answer modalities concerning activities such as standing up from a chair or carrying a weight. Each question has 3 response modalities: "No difficulty - 0 points" "a little - 1 point" or "a lot, unable - 2 points". A score > 4 indicates a risk of sarcopenia
  the kinematic parameters of the knee are measured via the Xsens sensors
percentage association of knee kinematics parameters with SARC-F score at 12 months | at 12 months
  evaluate the percentage of association between kinematic parameters and the SARC-F (Strength, assistance with walking, rising from a chair, climbing stairs, and falls) score
  SARC-F is for the early detection of sarcopenia. It contains 5 questions with 3 answer modalities concerning activities such as standing up from a chair or carrying a weight. Each question has 3 response modalities: "No difficulty - 0 points" "a little - 1 point" or "a lot, unable - 2 points". A score > 4 indicates a risk of sarcopenia
  the kinematic parameters of the knee are measured via the Xsens sensors
percentage association of knee kinematics with contractile function of the quadriceps at baseline | at baseline
  evaluate the percentage of association between kinematic parameters and contractile function of the quadriceps
  Measurement of isokinetic parameters on evaluation of the deficit on the healthy side/injured side with the ratio Quadriceps / Hamstrings
  the kinematic parameters of the knee are measured via the Xsens sensors
percentage association of knee kinematics with contractile function of the quadriceps at 12 months | at 12 months
  evaluate the percentage of association between kinematic parameters and contractile function of the quadriceps
  Measurement of isokinetic parameters on evaluation of the deficit on the healthy side/injured side with the ratio Quadriceps / Hamstrings
  the kinematic parameters of the knee are measured via the Xsens sensors
percentage association of knee kinematics parameters with body composition at baseline | at baseline
  evaluate the percentage of association between kinematic parameters and body composition
  Measurement of total body composition: appendicular lean mass (sum of lean mass of all 4 limbs: ALM) / height²); percentage of lean mass, visceral fat and whole body fat.
  the kinematic parameters of the knee are measured via the Xsens sensors
percentage association of knee kinematics parameters with body composition at at 12 months | at 12 months
  evaluate the percentage of association between kinematic parameters and body composition
  Measurement of total body composition: appendicular lean mass (sum of lean mass of all 4 limbs: ALM) / height²); percentage of lean mass, visceral fat and whole body fat.
  the kinematic parameters of the knee are measured via the Xsens sensors
percentage association of knee kinematics parameters with muscle mass at baseline | at baseline
  evaluate the percentage of association between kinematic parameters and muscle mass
  Measurement of muscle volume of both quadriceps and comparison of muscle changes between osteoarthritic and non-osteoarthritic knees.
  the kinematic parameters of the knee are measured via the Xsens sensors
percentage association of knee kinematics parameters with the biological function of muscle and joint cells at baseline | at baseline
  evaluate the percentage of association between kinematic parameters and the biological function of muscle and joint cells
  Measurement of the cross-sectional area of quadriceps muscle fibers. the kinematic parameters of the knee are measured via the Xsens sensors
percentage association of knee kinematics parameters with the number and size of myoblasts at baseline | at baseline
  evaluate the percentage of association between kinematic parameters and the biological function of muscle and joint cells
  Number and size of myoblasts obtained per satellite cell cultured on a longitudinal groove microstructured support.
  the kinematic parameters of the knee are measured via the Xsens sensors
percentage association of knee kinematics parameters with the differentiation capacity of mesenchymal stromal cells at baseline | at baseline
  evaluate the percentage of association between kinematic parameters and the biological function of muscle and joint cells
  Capacity of mesenchymal stromal cells (MSC) to differentiate into chondrocytes. the kinematic parameters of the knee are measured via the Xsens sensors
percentage association of knee kinematics with the senescence of musculoskeletal tissues at baseline | at baseline
  evaluate the percentage of association between kinematic parameters and the biological function of muscle and joint cells
  Measurement of the senescence of musculoskeletal tissues (chondrocytes, synoviocytes, adipocytes).
  the kinematic parameters of the knee are measured via the Xsens sensors

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Montpellier, Montpellier, France